CLINICAL TRIAL: NCT02729207
Title: A Phase II, Randomized, Double-blind, Placebo Controlled, Proof of Concept Study to Investigate the Safety and Efficacy of the Esflurbiprofen Hydrogel Patch in Treatment of Acute Pain Associated With Ankle Injury
Brief Title: Proof-of-concept Study of NSAID Hydrogel Patch in Treatment of Acute Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of patients number
Sponsor: Teikoku Seiyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TS-TK-254-US0200
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Ankle Sprain
Keywords: NSAID Patch
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esflurbiprofen 1.5% Hydrogel Patch (Active Comparator): One patch per 24hr for 7 days
  Interventions: Drug: Esflurbiprofen Hydrogel Patch
- Placebo comparator (Placebo Comparator): Placebo One patch per 24hr for 7 days
  Interventions: Drug: Esflurbiprofen Hydrogel Patch

INTERVENTIONS:
Drug: Esflurbiprofen Hydrogel Patch — One patch per day for 7 days

SUMMARY:
The safety and the efficacy of the Esflurbiprofen Hydrogel Patch will be assessed in comparing with placebo in the treatment of acute pain due to ankle sprain

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be a male or female aged 18 to 65 years, inclusive.
2. Subject must have a diagnosis of uncomplicated acute minor ankle sprain of Grade I or II as defined by the AAOS criteria.
3. Ankle sprain must have occurred <48 hours prior to Screening.
4. Subject must have a baseline self-evaluated pain score of >50 mm on a 100 mm VAS while bearing weight on the affected ankle.
5. Female subjects of childbearing potential must have a negative serum pregnancy test at Screening and be willing to use an acceptable form of birth control from the day of the first dose administration to 30 days after the last administration of the study product.
6. Subject must be willing to refrain from using any other pain medication (other than allowed rescue medication) during their participation.

Exclusion Criteria:

1. Subject is a pregnant, breastfeeding, or lactating female.
2. Subject has an acute ankle sprain of Grade III as defined by AAOS criteria.
3. Subject has an ankle fracture as confirmed by X-ray.
4. Ankle sprain requires surgical treatment.
5. Subject has experienced recurrent sprains (≥3 sprains of the same joint) or has sprained the affected joint within the last 12 months.
6. Subject has taken analgesics other than NSAID(s) or acetaminophen for any purpose within 7 days of Screening.
7. Subject has taken flurbiprofen or naproxen within 24 hours of Screening.
8. Ankle sprain is treated prior to Screening by ultrasound, physical therapy, or acupuncture.
9. Subject has used immunomodulators or immunosuppressive therapies (e.g., interferon, oral or parenteral corticosteroids, and cytotoxic drugs) within 4 weeks prior to randomization.
10. Subject has used any medicated topical agents (e.g., medicated creams or lotions) on the affected ankle within 7 days prior to Screening.
11. Subject is currently using any other medications that, in the opinion of the Investigator, may exacerbate or mask the anticipated side effects of NSAIDs or interfere with the Investigator's ability to monitor for them (e.g., blood thinners or proton-pump inhibitors).
12. Subject has non-intact or damaged skin in the area to be treated (e.g., eczema, psoriasis, exudative dermatitis, infected lesion, burn, or wound).
13. Subject has a history of ulcers, GI bleeding, hypertension, edema, heart failure, or CV disease.
14. Subject has asthma (except childhood asthma), urticaria, angioedema, or bronchospasm.

    a.A subject is eligible for the study if they have had no symptoms of these conditions that required medication in the 5 years prior to Screening.
15. Subject has a history of any chronic pain disorder.
16. Subject has coagulation defects.
17. Subject has a history of severe cardiac, renal, or hepatic impairment within 12 months prior to Screening that, in the opinion of the Investigator, would interfere with the outcome of the study.
18. Subject has a severe systemic disease (e.g., cancer or severe acute infection).
19. Subject has a known allergy or hypersensitivity to flurbiprofen, aspirin, other NSAID(s), or any excipient in the IP.
20. Subject has any systemic or dermatologic disorder that, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs.
21. Subject has a history of uncontrolled chronic or acute concomitant disease that, in the Investigator's opinion, would contraindicate study participation or confound interpretation of the results.
22. Subject has applied ice or compression to the affected ankle within 2 hours prior to Screening.
23. Subject has a bilateral ankle injury.
24. Subject has an ipsilateral knee injury. In the opinion of the Investigator, are unsuitable for inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-27 (Actual)

PRIMARY OUTCOMES:
Sum of intensity of pain difference after 48hr treatment (SPID48h) | 48hr after treatment starting
  SPID48h will be compared between EFHP and placebo.

SECONDARY OUTCOMES:
SPID24h | 24hr after treatment starting
  Sum of intensity (VAS) of pain difference after 24hr

OTHER OUTCOMES:
SPID72h | 72hr after treatment starting
  Sum of intensity (VAS) of pain difference after 72hr was measured

CONTACTS AND LOCATIONS:
Overall Officials: Masaru Kaneko, MD, Principal Investigator — SNBL Clinical Pharmacology Center
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No